CLINICAL TRIAL: NCT00506298
Title: A Randomized, Multi-Center Study to Compare the Effects of CRx-401 to Bezafibrate Plus Placebo on Plasma Glucose Levels When Given to Subjects With Type II Diabetes on Metformin.
Brief Title: Study of CRx-401 on Glucose Levels in Subjects With Type II Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zalicus (Industry)
Responsible Party: Medical Monitor, CombinatoRx
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRx-401-001
Record Dates: First submitted 2007-07-20; First posted 2007-07-25 (Estimated); Last update posted 2009-05-13 (Estimated); Status verified 2009-05

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; CRx-401; Bezafibrate; Diflunisal; Metformin; plasma glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Bezafibrate; Diflunisal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): CRx-401 (bezafibrate + diflunisal)
  Interventions: Drug: bezafibrate + diflunisal
- B (Active Comparator): bezafibrate + placebo
  Interventions: Drug: bezafibrate + placebo

INTERVENTIONS:
Drug: bezafibrate + diflunisal — bezafibrate + diflunisal
  Arms: A
Drug: bezafibrate + placebo — bezafibrate + placebo
  Arms: B

SUMMARY:
This trial will assess the efficacy of CRx-401 in lowering FPG levels in patients taking metformin to treat their diabetes. In addition, this initial trial will evaluate insulin resistance (HOMA-IR index), HgbA1c levels, glycated protein, LDL, HDL, triglycerides, and total cholesterol, as well as the safety of CRx-401.

ELIGIBILITY:
Inclusion Criteria:

* Must voluntarily give written informed consent
* Must be between 18-75 years of age
* Must have Type 2 diabetes for ≥ 6 months
* HgbA1C between 7.0% and 9.5%
* FPG > 6.7 mmol/L (120 mg/dL)
* BMI: Lower limit of 27 kg/m2 and an upper Limit of 45 kg/m2
* Treatment with a stable dosage for ≥ 8 weeks of either Glucophage metformin) ≥ 1000 and ≤ 2500 mg/day OR Glucophage XR ≤ 2000 mg/day
* eGFR ≥ 70 mL/min

Exclusion Criteria:

* History of any clinically significant atherosclerotic disorder including myocardial infarction (within 6 months of screening), angina, stroke, peripheral vascular disease or congestive heart failure
* Known hypersensitivity or idiosyncratic reaction related to fibrates or NSAIDs including photo-allergic or phototoxic reactions to fibrates
* Subjects in whom acute asthmatic attacks, urticaria, or rhinitis are precipitated by aspirin or other NSAIDs
* History of clinically significant (as determined by the investigator cardiac, hematologic, hepatobiliary, peptic ulcer, renal, immunologic, metabolic, urologic, pulmonary, endocrinologic, neurologic, dermatologic, psychiatric, and/or other major disease
* Type 1 Diabetes
* Evidence of Cushing's syndrome, untreated hypothyroidism or other disorders that may lead to secondary weight gain, insulin resistance, or Type 2 diabetes
* Proliferative diabetic retinopathy or significant neuropathic symptoms that also limit activities of daily living
* History of malignancy (except for treated or excised basal cell carcinoma)
* Surgery within the 90 days prior to screening except for minor dental or cosmetic procedures
* History of drug or alcohol abuse (as defined by the Investigator)
* History of opportunistic infection
* Serious local infection (e.g., cellulitis, abscess) or systemic infection (e.g., septicemia) within 3 months prior to screening
* Fever or symptomatic viral or bacterial infection within 2 weeks prior to screening
* Positive for HCV antibody
* Positive for HBsAg
* Known positive for HIV antibody
* Pharmacologic treatment with statins, unless dosage has been stable ≥ three months and is unlikely to change over the course of the study.
* Treatment with any concomitant medication that has not been at a stable dose for at least 28 days prior to screening.
* Currently taking or planning to take during the trial:

Sulphonylureas, Injected hypoglycemic (exanatide or insulin), Weight loss medications, Thiazolidenediones, Glucocorticoids (inhaled glucocorticoids are permitted), Digoxin, Anticoagulants, Phenytoin, Loratadine, Erythromycin, MAO-inhibitors, NSAIDs (ASA ≤ 81 mg/d is permitted), COX-2 Inhibitors, Cholestryramine or fibrates, DPP-IV inhibitors, Any herbal medications unless reviewed with study doctor

* Alanine aminotransferase ALT) or aspartate aminotransferase (AST laboratory values that exceed > 2.0 x upper limit of normal (ULN)
* White blood cell (WBC) count < 4.0 x 109 /L or >14.0 X 109 /L
* Hemoglobin < 105 g/L in females and < 110 g/L in males (< 10.5 g/dL in females and < 11.0 g/dL in males)
* Participation in another clinical trial and/or treatment received with any investigational agent within 30 days before the initial dose of study medication
* Female subject who is pregnant or lactating or of child bearing potential and not using acceptable methods of contraception (birth control pills, barriers or abstinence)
* Unwilling or unable to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the subject's return for follow-up visits on schedule
* Other unspecified reasons that, in the opinion of the Investigator or sponsor make the subject unsuitable for enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint will measure change in fasting plasma glucose from Baseline to Day 90 | Day 90

SECONDARY OUTCOMES:
The exploratory efficacy endpoints will measure change in the following parameters: HOMA Index, HgbA1C, fructosamine, LDL, HDL, OGTT, triglycerides and total cholesterol from Baseline to Day 90 | Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Tim Zmijowskyj, MD, Principal Investigator — Medicor Research Inc.
Locations (18):
- Canada (18):
  - Chilliwack, British Columbia
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Bay Roberts, Newfoundland and Labrador
  - Holyroad, Newfoundland and Labrador
  - St. John's, Newfoundland and Labrador
  - Aylmer, Ontario
  - Burlington, Ontario
  - Collingwood, Ontario
  - Corunna, Ontario
  - Greater Sudbury, Ontario
  - Robarts Research Institute, London, Ontario
  - London, Ontario
  - Newmarket, Ontario
  - Sarnia, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Saskatoon, Saskatchewan